CLINICAL TRIAL: NCT00034047
Title: Endometriosis : Traditional Medicine vs Hormone Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000453-01 (NIH)
Record Dates: First submitted 2002-04-19; First posted 2002-04-22 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Endometriosis; Pelvic pain; Acupuncture; Chinese herbs; Hormone therapy; Nafarelin
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Acupuncture Therapy; Nafarelin

INTERVENTIONS:
Procedure: Acupuncture
Drug: Chinese Products
Drug: Nafarelin

SUMMARY:
This 36-week study will determine whether traditional Chinese medicine (acupuncture and Chinese herbs) is as effective as hormone therapy for alleviating endometriosis-related pelvic pain.

DETAILED DESCRIPTION:
Endometriosis is a significant public health problem affecting 10-15% of women of childbearing age, many of whom suffer persistent pelvic pain and infertility. Therapeutic options include surgery and hormone therapy that are often temporarily effective but produce unwanted side-effects. The present proposal, based on case series reports of the effectiveness of Traditional Chinese Medicine (TCM: acupuncture and Chinese herbs) for this condition, aims to evaluate whether TCM is as effective as hormone therapy for alleviating endometriosis-related chronic pain.

Women with laparoscopy-diagnosed endometriosis will be randomly assigned to either TCM or hormone therapy. Women assigned to TCM will be divided into four sub-groups on the basis of the diagnostic categories of endometriosis recognized by TCM. A pre-established acupuncture protocol and herbal formula specific for each sub-group will be followed. This aspect of the research design permits an important feature of the clinical practice of TCM (matching treatment to sub-group diagnosis) to be adopted in a clinical trial. Women assigned to hormone therapy will be treated with the gonadotropin releasing hormone agonist (GnRHa), nafarelin, chosen for this study on the basis of its clinical trial-established efficacy, ease of patient usage via intranasal spray and milder side-effect profile relative to other GnRHa's. Pelvic pain symptoms (patient-scored) and signs (physician-scored) will be assessed at baseline, after 12 weeks of treatment, and at 12- and 24-week post-treatment follow-up. Pelvic examination scores will be determined by a physician blinded to the treatment group assignments. Side effects, including those of pseudomenopause known to result from GnRHa therapy, will be recorded in both groups at 4-week intervals during the 12-week treatment, and at each follow-up time. A further objective is to make a preliminary assessment of whether diagnostic sub-groups of endometriosis recognized by TCM serve as predictors of differential response to hormone therapy. Data obtained from this study, on treatment effectiveness, side effect profiles, recurrence of symptoms, compliance with therapy and drop-out rates, will be used to design a large-scale clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Women with laparoscopy-confirmed endometriosis within the past 6 years
* Experiencing chronic pelvic pain, dysmenorrhea (painful periods) and dyspareunia (painful intercourse), at least one of which is moderate to severe

Exclusion Criteria:

* Use of traditional Chinese medicine for endometriosis. If previous treatment with hormone therapy, must have responded positively but not have been on hormone therapy within the past 6 months
* Use of any form of hormone-based contraception during the 12-week treatment and 24-week follow-up periods
* Diagnosed with any chronic condition other than endometriosis, or any other acute condition that causes pain
* Pregnancy or breast feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Pain assessments

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hammerschlag, PhD, Principal Investigator — Oregon College of Oriental Medicine; Kenneth Burry, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health Sciences University, Women's Health Research Unit, Portland, Oregon
  - Oregon College of Oriental Medicine Clinic, Portland, Oregon